CLINICAL TRIAL: NCT00770926
Title: Physical Activity and Diet to to Reduce Disparities in Diabetes Risk
Brief Title: Reducing Disparities in Diabetes Risk Through Lifestyle Changes in Community Settings
Acronym: LWBW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R18DK067896-01A2 (NIH); R18DK067896 (NIH)
Record Dates: First submitted 2008-10-08; First posted 2008-10-10 (Estimated); Last update posted 2013-05-21 (Estimated); Status verified 2013-05

CONDITIONS: Diabetes
Keywords: risk reduction; minority; diabetes prevention; lifestyle program; behavior change
MeSH Terms: conditions — Diabetes Mellitus; Risk Reduction Behavior

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Program immediately (Experimental): Receives the lifestyle program as soon as possible after randomization
  Interventions: Behavioral: Live Well, Be Well
- Wait list control (No Intervention): Wait one year and at the end of the year, is offered the option of participating in the program

INTERVENTIONS:
Behavioral: Live Well, Be Well — Lifestyle change program using personal contact and telephone counseling
  Arms: Program immediately

SUMMARY:
This study aims to design and test the effectiveness of a lifestyle diabetes risk reduction program, Live Well, Be Well, in reducing risk of diabetes in persons at risk with a focus on reaching lower-income, minority individuals.

DETAILED DESCRIPTION:
To design and test the effectiveness of a lifestyle diabetes risk reduction program, Live Well, Be Well, to increase physical activity, decrease weight, and improve diet, offered in community-based settings to primarily lower income, minority persons aged 25 and older at moderate to high risk of diabetes. The design is a randomized controlled trial with the primary outcome being fasting plasma glucose; secondary outcomes are weight, physical activity, blood pressure, and other physiological risk factors as well as health-related quality of life. This project is a partnership between the University of California San Francisco and the City of Berkeley Division of Public Health.

ELIGIBILITY:
Inclusion Criteria:

* age 25 and older
* moderate- to high-risk score on a Diabetes Risk Appraisal (DRA) (assessing sedentary behavior, family history of diabetes, race/ethnicity, gestational diabetes, hypertension, and high cholesterol) and a fasting fingerstick glucose level of 95-140 mg/dL (indicating high risk of diabetes).
* conversant in English or Spanish

Exclusion Criteria:

1. diabetes, assessed by self-report of having ever been told by a physician that they have diabetes (other than gestational) OR use of an oral hypoglycemic medication or insulin, OR a fingerstick fasting glucose level of >150 mg/dl;
2. unstable chronic or serious condition that could limit participation in unsupervised light to moderate physical activity (e.g. unstable angina, diagnosed with or hospitalized for chest pain, heart surgery, stroke, or myocardial infarction in the past 6 months);
3. uncontrolled hypertension (systolic >180 mmHg or diastolic >105 mmHg);
4. current pregnancy or attempting to conceive;
5. plans to move from the area within 1 year;
6. insufficient cognitive functioning to complete program procedures,
7. implanted defibrillator,
8. a hip or knee replacement in the past 3 months.

Min Age: 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 230 (Actual)
Dates: Start 2006-09; Primary Completion 2009-08 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Body weight | one year

SECONDARY OUTCOMES:
diet | One year

CONTACTS AND LOCATIONS:
Overall Officials: Anita L Stewart, Ph.D, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco, San Francisco, California, United States

REFERENCES:
- [Result] Delgadillo AT, Grossman M, Santoyo-Olsson J, Gallegos-Jackson E, Kanaya AM, Stewart AL. Description of an academic community partnership lifestyle program for lower income minority adults at risk for diabetes. Diabetes Educ. 2010 Jul-Aug;36(4):640-50. doi: 10.1177/0145721710374368. Epub 2010 Jun 24. PMID 20576836
- [Result] Santoyo-Olsson J, Cabrera J, Freyre R, Grossman M, Alvarez N, Mathur D, Guerrero M, Delgadillo AT, Kanaya AM, Stewart AL. An innovative multiphased strategy to recruit underserved adults into a randomized trial of a community-based diabetes risk reduction program. Gerontologist. 2011 Jun;51 Suppl 1(Suppl 1):S82-93. doi: 10.1093/geront/gnr026. PMID 21565823